CLINICAL TRIAL: NCT04840550
Title: A Phase 3, Randomized, Double-blind, Active-controlled, Multicenter Study to Evaluate the Safety and Efficacy of Tegoprazan 25 mg for the Prevention of Peptic Ulcer Disease in Patients on Continuous Long-term Treatment With NSAIDs
Brief Title: Study to Evaluate the Safety, Efficacy of Tegoprazan for the Prevention of PUD in Patients on Treatment With NSAIDs
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: HK inno.N Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IN_APA_308
Record Dates: First submitted 2021-04-07; First posted 2021-04-12 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-01

CONDITIONS: Preventive Peptic Ulcer
MeSH Terms: interventions — Lansoprazole; tegoprazan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tegoprazan 25mg (Experimental): Tegoprazan 25mg tablets will be orally administered once a day, with NSAIDs, for up to 6 months.
  Interventions: Drug: Tegoprazan 25 mg
- Lansoprazole 15mg (Active Comparator): Lansoprazole 15mg capsules will be orally administered, once a day, with NSAIDs, for up to 6 months.
  Interventions: Drug: Lansoprazole 15 mg

INTERVENTIONS:
Drug: Lansoprazole 15 mg — Lansoprazole 15 mg tablets will be orally administered once a day, with NSAIDs, for up to 6 months.
  Arms: Lansoprazole 15mg
Drug: Tegoprazan 25 mg — Tegoprazan 25 mg tablets will be orally administered once a day, with NSAIDs, for up to 6 months.
  Arms: Tegoprazan 25mg

SUMMARY:
This study is designed to confirm the non-inferiority of Tegoprazan 25 mg, compared to Lansoprazole 15 mg, to prevent gastroduodenal ulcers and verify the safety of tegoprazan following oral administration of tegoprazan 25 mg QD or lansoprazole 15 mg QD in patients on long-term treatment with NSAIDs.

DETAILED DESCRIPTION:
This is a double-blind, randomized, active-controlled, phase 3 study. Subjects will be randomly assigned to one of the two treatment groups (tegoprazan 25 mg, lansoprazole 15 mg).

ELIGIBILITY:
Inclusion Criteria:

* ≥60 years of age, or ≥20 years of age with a history of gastroduodenal ulcers (gastric and/or duodenal ulcers) at screening
* Requires continued treatment with NSAIDs for ≥24 weeks

Exclusion Criteria:

* Has an active stage (A1, A2) or healing stage (H1, H2) of gastroduodenal ulcers per the Sakita-Miwa classification identified by upper GI endoscopy at screening
* Has uncontrolled severe hypertension
* Has severe heart failure, congestive heart failure (NYHA Ⅱ to Ⅳ), ischemic heart disease (unstable angina, myocardial infarction), or peripheral artery disease, or has undergone coronary artery bypass graft (CABG) who is considered ineligible for treatment with NSAIDs
* Has a positive H. pylori test at screening

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 390 (Estimated)
Dates: Start 2021-05-07 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects with gastric and/or duodenal ulcers at Week 24 | week 24
  The proportion of subjects with gastric and/or duodenal ulcers on upper GI endoscopy at Week 24

SECONDARY OUTCOMES:
Proportion of subjects without NSAID-related GI symptoms at Weeks 4, 12, and 24 | week 4, 12, 24
  GI symptoms are as follows; Heartburn, Regurgitation, Upper abdominal pain or discomfort

CONTACTS AND LOCATIONS:
Overall Officials: Jea Jun Kim, Principal Investigator — Samsung Medical Center
Locations (2):
- South Korea (2):
  - Samsung Medical Center, Seoul
  - The catholic univ. of Korea Eunpyeong ST. Mari's hospital, Seoul

IPD SHARING:
Plan to Share IPD: No